CLINICAL TRIAL: NCT02591628
Title: Treatment of Hypertension In Adults With ThiaZIDES: Pragmatic Trial Pilot Study
Acronym: ThiaZIDES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34HL119790 (NIH)
Record Dates: First submitted 2015-09-25; First posted 2015-10-29 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-01

CONDITIONS: Hypertension
Keywords: Hypertension; Thiazide diuretics
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Intervention is HCTZ prescription conversion to chlorthalidone. Intervention patients are defined as patients of physicians randomized to "intervention." All these patients will have their current prescription of hydrochlorothiazide (HCTZ) switched to an equipotent dose of Chlorthalidone. These patients can choose to decline this intervention, and will be followed for 9 months with no other intervention to observe primary and secondary outcomes.
  Interventions: Behavioral: HCTZ prescription conversion to chlorthalidone
- Usual Care (No Intervention): Usual care patients are defined as patients of physicians randomized to "usual care." All these patients will keep their current prescription for HCTZ and work with their physician like normal. These patients will be followed for 9 months with no intervention to compare primary and secondary outcomes to the intervention group.

INTERVENTIONS:
Behavioral: HCTZ prescription conversion to chlorthalidone — The intervention is simply a prescription conversion and the main outcome is whether or not patients accept the conversion and treatment with chlorthalidone.
  Arms: Intervention

SUMMARY:
This proposed pilot study will test methods and feasibility for a large pragmatic clinical trial comparing two inexpensive, first-line drugs for treating high blood pressure to determine if one is superior in preventing serious cardiovascular events and death. It will develop and test novel approaches to conducting trials that will be faster, less expensive, and more realistic by being embedded in a typical practice setting and using advanced health information technology.

DETAILED DESCRIPTION:
For several decades, U.S. hypertension treatment guidelines have recommended a low-dose diuretic such as hydrochlorothiazide (HCTZ) or chlorthalidone (CTD) as initial monotherapy in a stepped-care approach or as part of an initial two-drug combination. In numerous large clinical trials, CTD-based regimens have significantly reduced rates of cardiovascular events such as stroke, heart failure, and cardiovascular mortality compared with placebo, usual care, or active comparators. In contrast, few outcome studies have compared HCTZ-based regimens with other treatments, and they have generally found HCTZ to be less effective than non-thiazide comparators in preventing cardiovascular events. The two drugs have never been compared directly in a large trial. Despite the empirical evidence favoring CTD, HCTZ is much more widely used in clinical practice. The proposed R34 is a pilot study conducted in two large integrated health systems to test methods and feasibility for an eventual pragmatic randomized trial comparing the effectiveness of HCTZ and CTD for preventing cardiovascular events and mortality. Using a cluster-randomized design, investigators will allocate 40 primary care physicians and their adult hypertensive patients who currently use HCTZ (N=2,000) to either convert HCTZ users to CTD (intervention group) or to continue HCTZ (usual care group). The pilot study and planned full-scale trial will use existing health care infrastructure and electronic health records to identify eligible study subjects, distribute study medication, and collect operational and outcomes data. For this pilot study, Aim 1 will document that the intervention is delivered as intended. Aim 2 will compare safety in intervention and usual care patients. Aim 3 will refine the pilot study design and identify critical factors for intervention success using a mixed-methods approach. Aim 4 will refine estimates of sample size. Finally, Aim 5 will determine the costs of ascertaining outcomes and estimate per-participant costs for the full-scale trial. The pilot study will produce data that are necessary and sufficient to inform the planning of a full-scale trial comparing CTD and CTZ and will advance the development of methods for pragmatic trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older
* Hypertension diagnosis (ICD-9 401.x)
* Current prescription for hydrochlorothiazide (HCTZ), 12.5-50 mg/day as a single-agent (not part of a fixed-dose combination drug)
* No history of intolerance to chlorthalidone (CTD)
* No known low levels of sodium (<135 mEg/L (milliequivalents per liter)) or potassium (<3.5 mEg/L)
* English speaking

Exclusion Criteria:

* Physician deems patient inappropriate for switching HCTZ to CTD
* Patient refuses the switch prior to intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2027 (Actual)
Dates: Start 2015-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Conversion to chlorthalidone, number of patients with primary fills | 3 months
  We will observe pharmacy claims to assess whether intervention patients filled their first prescription for chlorthalidone (primary adherence)
Conversion to chlorthalidone, number of participants with secondary fills | 9 months
  We will observe pharmacy claims to assess whether intervention patients who filled their first chlorthalidone prescription also filled their subsequent prescription (secondary adherence)

SECONDARY OUTCOMES:
Blood pressure | 9 months
  Systolic and diastolic blood pressure measures, as documented in electronic health record
Hypertension drugs | 9 months
  Use of anti-hypertensive drugs in addition to hydrochlorothiazide or chlorthalidone, as documented in pharmaceutical claims
Electrolyte levels | 9 months
  Sodium and potassium levels, as documented in electronic health record
Renal function | 9 months
  Kidney function lab values (including epidermal growth factor receptor (eGFR) and creatinine), as documented in electronic health record
Safety outcomes | 9 months
  Hypotension with fainting (over-treatment), hypertensive crisis (under-treatment) and other clinical outcomes related to safety of hypertension treatment

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Margolis, MD, MPH, Principal Investigator — HealthPartners Institute; Stephen P Fortmann, MD, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - HealthPartners Institute for Education and Research, Bloomington, Minnesota
  - Kaiser Permanente Center for Health Research, Portland, Oregon